CLINICAL TRIAL: NCT05260632
Title: Effect of Smartphone Addiction on Manual Coordination, Strength and Hand Pain in Normal Teenage Students
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Eid Mohamed Youssif, assistant lecturer, Cairo University
Other Study IDs: P.T.REC/012/003440
Record Dates: First submitted 2022-02-19; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Smart Phone Addiction, Manual Coordination, Hand Grip Strength, Pinch Strength, Teenage Students

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- no intervention
- 2 groups

SUMMARY:
Statement of the problem:

• Does addiction of smart phone affect upper limb coordination, manual dexterity, hand grip and pinch strength?

Null Hypotheses:

• Addiction of smart phone does not affect upper limb coordination, manual dexterity, hand grip and pinch strength in normal teenage students.

DETAILED DESCRIPTION:
Subjects:

The survey targets the normal teenage students from both sexes. Sample size estimation will be carried out to determine the recruited number of students, selected randomly from both governmental and private preparatory and secondary schools at Ashmoon educational administration, Menofia Governorate to participate in this study.

Study design:

Cross sectional observational study. Sample design will be a cluster sample,

A. Inclusion criteria:

1. The students' age will range from 12 to 18 years.
2. Normal students including both boys and girls.
3. Participants have a range score from 31 to 60 points for boys and from 33 to 60 points for girls on smartphone addiction scale according to Kwon et al (2013).
4. Their body mass index will be within the normal range according to WHO indices .
5. Cooperative students who wish to participate in the current study.
6. The students will represent different socioeconomic levels.

B. Exclusion criteria:

The students will be excluded from the study if they have one of the following:

1. Congenital abnormalities or medical conditions, which may affect the study.
2. Musculoskeletal problems such as previous or recent orthopedic surgery, fractures, prostheses, inflammation of the fingers, arms, or shoulder.
3. Visual or hearing defects.
4. Motor, behavioral, or neurologic disorders and learning disabilities. • Participants have a range score from 31 to 60 points for boys and from 33 to 60 points for girls on smartphone addiction scale, then participants will be divided into 2 levels of addiction.

Assessment of manual dexterity and upper extremity coordination will be carried out by using The Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2) (Bruininks and Bruininks, 2005). Hand grip strength and pinch strength will be assessed by hand dynamometer and pinch meter.

ELIGIBILITY:
Inclusion Criteria:

1. The students' age will range from 12 to 18 years.
2. Normal students including both boys and girls.
3. Participants have a range score from 31 to 60 points for boys and from 33 to 60 points for girls on smartphone addiction scale according to Kwon et al (2013).
4. Their body mass index will be within the normal range according to WHO indices .
5. Cooperative students who wish to participate in the current study.
6. The students will represent different socioeconomic levels.

Exclusion Criteria:

The students will be excluded from the study if they have one of the following:

1. Congenital abnormalities or medical conditions, which may affect the study.
2. Musculoskeletal problems such as previous or recent orthopedic surgery, fractures, prostheses, inflammation of the fingers, arms, or shoulder.
3. Visual or hearing defects.
4. Motor, behavioral, or neurologic disorders and learning disabilities

   -

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Assessment of Manual coordination | Baseline - one hour for each participant
  Assessment of change in manual dexterity and upper extremity coordination will be carried out by using The Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2) (Bruininks and Bruininks, 2005).
Assessment of hand grip strength | Baseline - one hour for each participant
  Assessment of change in Hand grip strength will be assessed by hand dynamometer device.
Assessment of pinch strength | Baseline - one hour for each participant
  Assessment of change in pinch strength by pinchmeter device.

CONTACTS AND LOCATIONS:
Overall Officials: Amira Mohamed, Principal Investigator — Cairo University
Locations (1):
- Outpatient clinic, Faculty of Physical Therapy, Cairo university, Cairo, Egypt